CLINICAL TRIAL: NCT00103623
Title: Incidence of Immediate Onset Systemic Allergic Reactions in Patients Treated With Plenaxis®
Brief Title: The Plenaxis® Experience Study
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: PRAECIS Pharmaceuticals Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 149-IV-01
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: Advanced; Symptomatic; Prostate; Cancer; Advanced Symptomatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — abarelix

INTERVENTIONS:
Drug: Plenaxis

SUMMARY:
Praecis is currently conducting a 2000 patient Experience Study; this is a Phase IV commitment postmarketing safety study in the Food and Drug Administration (FDA) indicated population of patients receiving Plenaxis®. The purpose of the study is to estimate the incidence of immediate-onset systemic allergic reactions in the indicated population receiving Plenaxis® and to determine whether the hazard rate changes over time.

DETAILED DESCRIPTION:
This is a postmarketing patient safety study in the FDA indicated population of patients receiving Plenaxis®. On a quarterly basis, patients enrolled in the Plenaxis® Experience Study will have their charts audited to record the number of immediate-onset systemic allergic reactions that may occur while receiving Plenaxis®. The study will close when 2,000 patients have been enrolled. If immediate onset allergic reactions occur, patients may be eligible to enroll in a second protocol (skin testing in patients who experience an immediate onset allergic reaction). Collection of all immediate-onset systemic allergic reactions will continue for each patient enrolled in the study until the patient discontinues Plenaxis® for any reason, the patient withdraws consent to continue in the study or the patient is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible to participate in the study if he meets the following criteria:

* Male ≥ 18 years old with advanced symptomatic prostate cancer for whom LHRH agonist therapy is not appropriate and who refuses surgical castration
* Has at least one of the following:

  1. Risk of neurological compromise due to metastases,
  2. Ureteral or bladder outlet obstruction due to local encroachment or metastatic disease or
  3. Severe bone pain from skeletal metastases persisting on narcotic analgesia
* Patients or their legal representatives must be able to read, understand and sign an informed consent form to participate in the trial.

Exclusion Criteria:

* Female Patients,
* Pediatric patients,
* Patients with known hypersensitivity to any of the components in the abarelix injectable suspension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2004-06; Study Completion 2008-12

PRIMARY OUTCOMES:
Estimate the incidence of immediate-onset systemic allergic reactions in the indicated population receiving Plenaxis

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Riedel, PhD, Study Director — PRAECIS Pharmaceuticals Inc.
Locations (60):
- United States (60):
  - Millenium Therapeutics & Research - Urology Practice, Birmingham, Alabama
  - Valley Urologic Associates, Goodyear, Arizona
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Arizona Urologic Specialists, Tucson, Arizona
  - Alfred Sidhom, MD, FACS, PC, Anaheim, California
  - Dr. Chris Threatt, Atherton, California
  - Hematology-Oncology Group of Fresno, Fresno, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - Atlantic Urological Medical Group, Long Beach, California
  - Paul Neustein, MD. INC, Poway, California
  - San Diego Urology, San Diego, California
  - Sherman Oaks Urological Medical Group, Inc., Sherman Oaks, California
  - Urology Associates PC, Denver, Colorado
  - Urologic Associates, Fort Meyers, Florida
  - Southwest Florida Urologic Associates, Fort Myers, Florida
  - University of Florida Shands Jacksonville, Jacksonville, Florida
  - UroSearch, Ocala, Florida
  - Urology Associates of Ocala, P.A., Ocala, Florida
  - South Florida Urology Center Inc, Pembroke Pines, Florida
  - South Florida Urology Center, Inc., Pembroke Pines, Florida
  - Uro-Medix, Inc, Sunrise, Florida
  - Osvaldo F. Padron MD, FACS, Tampa, Florida
  - Urological Surgical Services, Tavares, Florida
  - Osler Medical, West Melbourne, Florida
  - Urology Associates, P.C., Marietta, Georgia
  - Praire Medical Associates, LTD, Chicago, Illinois
  - Midwest Prostate Urology Health Center, Chicago, Illinois
  - Urology of Indiana, Indianapolis, Indiana
  - Unity HealthCare DBA Lafayette Clinic of Urology, Lafayette, Indiana
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Private Practice, Emporia, Kansas
  - KUMC Department of Urology, Kansas City, Kansas
  - Tri-County Urology, Milford, Massachusetts
  - Bay State Clinical Trials Inc, Watertown, Massachusetts
  - Lakeside Urology, Saint Joseph, Michigan
  - Tewodros Fresseha MD PC, Southfield, Michigan
  - Midwest Urology, Independence, Missouri
  - Kansas City Urology Care, Kansas City, Missouri
  - Quality Clinical Research, LLC, Omaha, Nebraska
  - Sheldon j. Freedman, MD Ltd, Las Vegas, Nevada
  - Essex-Hudson Urology, Bloomfield, New Jersey
  - Hunterdon Urological Associates, PA, Flemington, New Jersey
  - Northwest Urology Associates, Morristown, New Jersey
  - Roseland Surgical Suite, Roseland, New Jersey
  - Urology Healthcare Associates/Rancocas Medical Center, Willingboro, New Jersey
  - Staten Island Urological Research, PC, Staten Island, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - American Health Research, Charlotte, North Carolina
  - Northeast Urology Research, Concord, North Carolina
  - Washington Urological Associates, Washington, North Carolina
  - Columbus Urology Research, Columbus, Ohio
  - Parkhurst Research Organization, Bethany, Oklahoma
  - Bryn Mawr Urology, Devon, Pennsylvania
  - Dr. Peter Sinaiko, Langhorne, Pennsylvania
  - Urology and Urological Oncology, Philadelphia, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Dr. Greg Echt, Irving, Texas
  - North West Prostate Institute, Seattle, Washington
  - Roger D. Fincher, MD, Spokane, Washington